CLINICAL TRIAL: NCT01428271
Title: Comparison Between the Expected Site of Sacral Hiatus by Conventional Method and the Real Site by Ultrasonography for Caudal Block in Children
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2011-0337
Record Dates: First submitted 2011-08-10; First posted 2011-09-02 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Inguinal Herniorraphy
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Herniorrhapy with caudal block: Children aged 0-72 months who are scheduled to undergo elective inguinal herniorrhapy under general anesthesia with caudal block
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — The confirmation of the real site of the sacral hiatus by ultrasonography

SUMMARY:
Caudal block is one of the most useful and popular regional block in pediatric anesthetic practice. Successful caudal block depends on the proper placement of a needle through sacral hiatus by following anatomical landmarks. The sacrum and the position of sacral hiatus are extreme variable anatomical structure. Generally, the equilateral triangle located between the apex of the sacral hiatus and posterior superior iliac spines is used in determining the location of the sacral hiatus as the conventional method. Previous study demonstrated that the triangle formed between the apex of the sacral hiatus and the posterior superior iliac spines was found to have the features of an equilateral triangle in adult. There is no study about the efficacy of the conventional method using the equilateral triangle in children. In this study, the investigators will compare between the expected site of sacral hiatus by conventional method using the equilateral triangle and the real site of the sacral hiatus confirmed by ultrasonography for caudal block in children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-72 months
* patient whho are scheduled to undergo elective inguinal herniorraphy under general anesthesia

Exclusion Criteria:

* The history of prematurity
* he histories of the infection, tumor, and operation in sacrum 3. The history or suspicion of meningomyelocele

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged 0-72 months who are scheduled to undergo elective inguinal herniorraphy under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
the expected site of the sacral hiatus by convential method | approximately 5 minutes after general anesthesia
  1)The distance bewteen the midpoint of posterior superior iliac spines and the expected site of sacral hiatus by conventional method and 2)the distance between the midpoint of posterior superior iliac spines and the real site of sacral hiatus by ultrasonography.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Background] Senoglu N, Senoglu M, Oksuz H, Gumusalan Y, Yuksel KZ, Zencirci B, Ezberci M, Kizilkanat E. Landmarks of the sacral hiatus for caudal epidural block: an anatomical study. Br J Anaesth. 2005 Nov;95(5):692-5. doi: 10.1093/bja/aei236. Epub 2005 Sep 9. PMID 16155035